CLINICAL TRIAL: NCT00255034
Title: Phase IV Study of Tailored Therapy With Peg Interferon Alfa 2b and Ribavirin for Patients With Genotype 3 and High Viral Load. Genotype 3 Extended Treatment for HCV (GET-C Study)
Brief Title: Effects of 48 Weeks Versus 24 Weeks of Therapy With Peg-Intron/Ribavirin in Patients With Chronic Hepatitis C, Genotype 3 (Study P04143)(TERMINATED)
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Recruitment targets were unachievable in the currently available population.
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P04143
Record Dates: First submitted 2005-11-15; First posted 2005-11-17 (Estimated); Results first posted 2009-07-23 (Estimated); Last update posted 2017-04-06 (Actual); Status verified 2017-03

CONDITIONS: Hepatitis C, Chronic
Keywords: chronic hepatitis C; pegylated interferon alfa-2b; ribavirin; Australia
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — peginterferon alfa-2b; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 24 weeks of therapy (Active Comparator): Genotype 3 HCV subjects with high viral load (at least 2 million copies/mL) treated for 24 weeks
  Interventions: Biological: Peginterferon alfa-2b; Drug: Ribavirin
- 48 weeks of therapy (Experimental): Genotype 3 HCV subjects with high viral load (at least 2 million copies/mL) treated for 48 weeks
  Interventions: Biological: Peginterferon alfa-2b; Drug: Ribavirin

INTERVENTIONS:
Biological: Peginterferon alfa-2b — Powder for injection in Redipen (50, 80, 100, 120 and 150 microgram strengths), subcutaneous, dose of 1.5 micrograms/kg, weekly for up to 24 weeks
  Other Names: SCH 54031, PegIntron
  Arms: 24 weeks of therapy
Biological: Peginterferon alfa-2b — Powder for injection in Redipen (50, 80, 100, 120 and 150 microgram strengths), subcutaneous, dose of 1.5 micrograms/kg, weekly for up to 48 weeks
  Other Names: SCH 54031 PegIntron
  Arms: 48 weeks of therapy
Drug: Ribavirin — 200 mg capsules, oral, weight-based dose of 800, 1000, or 1200 mg, daily for up to 24 weeks
  Other Names: SCH 18908 Rebetol
  Arms: 24 weeks of therapy
Drug: Ribavirin — 200 mg capsules, oral, weight-based dose of 800, 1000, or 1200 mg, daily for up to 48 weeks
  Other Names: SCH 18908 Rebetol
  Arms: 48 weeks of therapy

SUMMARY:
This is an Australian, open-label, multicenter, randomized, double-blind clinical trial designed to assess the efficacy of combination therapy with pegylated interferon alfa-2b and ribavirin for 48 weeks versus 24 weeks in the treatment of chronic hepatitis C (treatment-naïve genotype 3 subjects with high viral loads who have a METAVIR score of at least F1A2). The primary endpoint will be a sustained virological response defined by undetectable HCV RNA in serum at 24 weeks after completion of therapy.

ELIGIBILITY:
Inclusion Criteria:

* Comply with all current Australian Schedule of Pharmaceutical Benefits S100 eligibility criteria.
* Chronic hepatitis C genotype 3 infection with a viral load of at least 2 million copies per mL.
* Able to give written informed consent.
* Understand and be able to adhere to the dosing and visit schedules.
* Compensated liver disease with the following minimum hematologic and biochemical criteria:

  * Hemoglobin ≥120 g/L (females), ≥130 g/L (males)
  * Platelets ≥100 x 10^9/L
  * Neutrophil count ≥1.5 x 10^9/L
  * Creatinine clearance >50 mL/minute
  * Thyroid stimulating hormone (TSH) within normal limits
* Serum hepatitis B surface antigen (HBsAg) and human immunodeficiency virus (HIV) negative.
* Negative pregnancy test.

Exclusion Criteria:

* Suspected hypersensitivity to interferon, pegylated interferon alfa-2b, or ribavirin.
* Participation in any other investigational drug program within 30 days of the screening visit for this protocol.
* Any cause of liver disease based on patient history and biopsy other than chronic hepatitis C, including but not limited to: hemochromatosis, alpha-1 antitrypsin deficiency, Wilson's disease, autoimmune hepatitis, alcoholic liver disease, drug-related liver disease.
* Hepatocellular carcinoma.
* Decompensated cirrhosis (ascites, history of encephalopathy or bleeding varices, serum albumin <35 g/L, prothrombin time (PT) prolonged by greater than 3 sec).
* Significant cardiovascular dysfunction within the past 6 months (e.g., angina, congestive heart failure, myocardial infarction, severe hypertension, or significant arrhythmia) or participants with an ECG showing clinically significant abnormalities.
* Immunologically-mediated disease, (e.g. inflammatory bowel disease), idiopathic thrombocytopenic purpura, systemic lupus erythematosus, autoimmune hemolytic anemia, scleroderma, severe psoriasis).
* Hemophilia or any hemoglobinopathy, including but not limited to thalassemia major.
* Severe psychiatric condition, including major depression, a history of major psychoses, current suicidal ideation, and/or suicidal attempts.
* Ongoing substance abuse, e.g. alcohol, I.V. drugs or inhalants that in the opinion of the investigator would jeopardize the patient's ability to comply with study requirements.
* Clinically significant ophthalmological disorders.
* Treatment or recent treatment with immunosuppressive agents (excluding short-term corticosteroid withdrawal) and immunosuppressed transplant recipients.
* Poorly controlled thyroid disease.
* Any other condition that in the opinion of the investigator would make the patient unsuitable for enrolment, or could interfere with the patient participating in and completing the clinical trial program.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2005-02; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The target recruitment was not attained within the anticipated study time-frame and so study recruitment was ceased on 24 November 2006; however those patients already enrolled in the study continued in the study until completion.
Pre-assignment Details: Enrolled 146 subjects; 143 subjects were treated; 3 subjects were withdrawn at Baseline and never received study medication: 1 subject in the 24 weeks group due to consent issues; and 2 subjects in the 48 weeks group (1 subject was ineligible and 1 subject was randomized in error).
Period: Overall Study
Arm/Group | 24 Weeks of Therapy | 48 Weeks of Therapy
Started | 79 | 64
Completed | 64 | 26
Not Completed | 15 | 38
Not completed — Withdrawal by Subject | 15 | 38

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 24 Weeks of Therapy | 48 Weeks of Therapy | Total
Number analyzed (Participants) | 79 | 64 | 143
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.9 (9.20) | 40.5 (9.80) | 40.7 (9.44)
Sex/Gender, Customized [Number; unit: participants]
  Female | 27 | 12 | 39
  Male | 52 | 51 | 103
  Transgender | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Sustained Virological Response (SVR), Defined by Undetectable HCV RNA in Serum at 24 Weeks After Completion of Therapy
Description: No formal comparisons could be made and no conclusions drawn because of small numbers in the treatment groups; a result of an inability to fulfill the recruitment target.
Time Frame: 24 weeks after completion of either up to 24 or 48 weeks of therapy
Population: Data were missing for 1 subject in the "48 weeks of therapy" treatment arm.
Measure: Number; unit: Participants
Arm/Group | 24 Weeks of Therapy | 48 Weeks of Therapy
Number analyzed (Participants) | 79 | 63
Participants | 55 | 36

ADVERSE EVENTS:
Arm/Group | 24 Weeks of Therapy | 48 Weeks of Therapy
Serious Adverse Events (participants affected / at risk) | 8/79 | 9/64
Other Adverse Events (participants affected / at risk) | 79/79 | 64/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 24 Weeks of Therapy (N=79) | 48 Weeks of Therapy (N=64)
NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
THYROIDITIS (Endocrine disorders) | 0 (0) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 (0) | 1 (2)
ASCITES (Gastrointestinal disorders) | 0 (0) | 1 (1)
INGUINAL HERNIA (Gastrointestinal disorders) | 0 (0) | 1 (1)
SALIVARY GLAND CALCULUS (Gastrointestinal disorders) | 1 (1) | 0 (0)
ABASIA (General disorders) | 1 (1) | 0 (0)
BUDD-CHIARI SYNDROME (Hepatobiliary disorders) | 0 (0) | 1 (1)
ABDOMINAL ABSCESS (Infections and infestations) | 1 (1) | 0 (0)
CELLULITIS (Infections and infestations) | 2 (2) | 0 (0)
MENINGITIS VIRAL (Infections and infestations) | 1 (1) | 0 (0)
SIALOADENITIS (Infections and infestations) | 1 (1) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0)
WOUND INFECTION (Infections and infestations) | 1 (1) | 0 (0)
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
NECK INJURY (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
DIZZINESS (Nervous system disorders) | 1 (2) | 0 (0)
SYNCOPE (Nervous system disorders) | 1 (1) | 0 (0)
TARDIVE DYSKINESIA (Nervous system disorders) | 1 (1) | 0 (0)
ANXIETY (Psychiatric disorders) | 1 (1) | 0 (0)
CONFUSIONAL STATE (Psychiatric disorders) | 1 (1) | 0 (0)
DELUSIONAL DISORDER, PERSECUTORY TYPE (Psychiatric disorders) | 0 (0) | 1 (1)
DEPRESSION (Psychiatric disorders) | 2 (2) | 0 (0)
HYPOMANIA (Psychiatric disorders) | 1 (1) | 0 (0)
SUICIDAL IDEATION (Psychiatric disorders) | 1 (1) | 0 (0)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
ECZEMA (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 24 Weeks of Therapy (N=79) | 48 Weeks of Therapy (N=64)
ANAEMIA (Blood and lymphatic system disorders) | 3 (3) | 5 (6)
NEUTROPENIA (Blood and lymphatic system disorders) | 2 (2) | 7 (9)
PALPITATIONS (Cardiac disorders) | 2 (2) | 4 (4)
DRY EYE (Eye disorders) | 2 (2) | 4 (4)
VISION BLURRED (Eye disorders) | 3 (3) | 7 (7)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 4 (4) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 4 (4) | 3 (3)
CHEILITIS (Gastrointestinal disorders) | 5 (6) | 2 (2)
CONSTIPATION (Gastrointestinal disorders) | 9 (10) | 5 (5)
DIARRHOEA (Gastrointestinal disorders) | 18 (18) | 8 (11)
DRY MOUTH (Gastrointestinal disorders) | 8 (8) | 5 (5)
MOUTH ULCERATION (Gastrointestinal disorders) | 6 (7) | 3 (3)
NAUSEA (Gastrointestinal disorders) | 28 (34) | 25 (27)
TOOTHACHE (Gastrointestinal disorders) | 3 (4) | 4 (4)
VOMITING (Gastrointestinal disorders) | 9 (13) | 6 (8)
CHEST PAIN (General disorders) | 0 (0) | 4 (4)
CHILLS (General disorders) | 13 (14) | 10 (10)
FATIGUE (General disorders) | 38 (40) | 30 (34)
INFLUENZA LIKE ILLNESS (General disorders) | 40 (40) | 41 (47)
INJECTION SITE ERYTHEMA (General disorders) | 15 (15) | 14 (14)
IRRITABILITY (General disorders) | 20 (24) | 20 (20)
PYREXIA (General disorders) | 7 (7) | 4 (4)
THIRST (General disorders) | 5 (5) | 1 (1)
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 (2) | 4 (4)
NASOPHARYNGITIS (Infections and infestations) | 7 (8) | 1 (1)
ORAL CANDIDIASIS (Infections and infestations) | 4 (4) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 6 (6) | 3 (3)
WEIGHT DECREASED (Investigations) | 6 (6) | 8 (9)
ANOREXIA (Metabolism and nutrition disorders) | 3 (3) | 4 (4)
DECREASED APPETITE (Metabolism and nutrition disorders) | 22 (26) | 14 (14)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 13 (14) | 9 (12)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 12 (13) | 12 (14)
MYALGIA (Musculoskeletal and connective tissue disorders) | 24 (31) | 12 (15)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 2 (2) | 6 (7)
DISTURBANCE IN ATTENTION (Nervous system disorders) | 7 (7) | 8 (9)
DIZZINESS (Nervous system disorders) | 8 (9) | 9 (11)
DYSGEUSIA (Nervous system disorders) | 5 (5) | 4 (4)
HEADACHE (Nervous system disorders) | 40 (51) | 34 (41)
LETHARGY (Nervous system disorders) | 18 (21) | 17 (20)
MEMORY IMPAIRMENT (Nervous system disorders) | 5 (5) | 4 (4)
ANXIETY (Psychiatric disorders) | 6 (6) | 10 (12)
DEPRESSED MOOD (Psychiatric disorders) | 5 (5) | 5 (6)
DEPRESSION (Psychiatric disorders) | 20 (21) | 17 (20)
INSOMNIA (Psychiatric disorders) | 30 (33) | 19 (21)
MOOD SWINGS (Psychiatric disorders) | 7 (7) | 10 (10)
SLEEP DISORDER (Psychiatric disorders) | 4 (4) | 10 (12)
COUGH (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 6 (6)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 15 (16) | 8 (9)
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (6)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 1 (1)
PHARYNGOLARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 5 (5)
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 0 (0)
ALOPECIA (Skin and subcutaneous tissue disorders) | 15 (16) | 11 (11)
DRY SKIN (Skin and subcutaneous tissue disorders) | 15 (15) | 9 (11)
ECZEMA (Skin and subcutaneous tissue disorders) | 3 (4) | 5 (5)
PRURITUS (Skin and subcutaneous tissue disorders) | 15 (17) | 10 (12)
RASH (Skin and subcutaneous tissue disorders) | 14 (15) | 16 (21)
RASH PRURITIC (Skin and subcutaneous tissue disorders) | 9 (12) | 3 (3)

LIMITATIONS AND CAVEATS:
No formal comparisons could be made and no conclusions drawn because of small numbers in the treatment groups; a result of an inability to fulfill the recruitment target.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less